CLINICAL TRIAL: NCT02811913
Title: Can rTMS Enhance Somatosensory Recovery After Stroke?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: N1767-P; 12025-H13 (Other: Louis Stokes Cleveland VA Medical Center IRB); NCT04535232 (obsolete NCT alias)
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: sensory impairment; sensory deficit; upper limb; transcranial magnetic stimulation; brain stimulation; rehabilitation
MeSH Terms: conditions — Stroke; Hypesthesia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High frequency rTMS (Other): Each subject is provided with three different brain stimulation interventions in a single arm, single session crossover design study. One of the sessions was 5 Hz rTMS
  Interventions: Other: repetitive transcranial magnetic stimulation (rTMS); Other: peripheral sensory stimulation
- Low frequency rTMS (Other): Each subject is provided with three different brain stimulation interventions in a single arm, single session crossover design study. One of the sessions was 1 Hz rTMS
  Interventions: Other: repetitive transcranial magnetic stimulation (rTMS); Other: peripheral sensory stimulation
- Sham rTMS (Other): Each subject is provided with three different brain stimulation interventions in a single arm, single session crossover design study. One of the sessions was sham rTMS
  Interventions: Other: repetitive transcranial magnetic stimulation (rTMS); Other: peripheral sensory stimulation

INTERVENTIONS:
Other: repetitive transcranial magnetic stimulation (rTMS) — 3 types of interventions on different sessions
  * session 1 - High frequency rTMS targeting contralesional sensory cortex
  * session 2 - Low frequency rTMS
  * session 3 - sham rTMS
Other: peripheral sensory stimulation — peripheral sensory electrical stimulation and vibration of the stroke-affected hand administered concurrently with each rTMS

SUMMARY:
Stroke affects over 795,000 Americans every year and has an enormous impact on the well-being of American Veterans with 6,000 new stroke admissions every year. Many of these stroke survivors are living with disabilities that limit their everyday function. One of the major consequences of stroke is loss of sensation which manifests as inability to perceive touch, temperature, pain or limb movement. Lack of sensation hinders full functional recovery. Current treatments for sensory loss produce only limited improvements and do not achieve full recovery. Therefore, it is critical to develop new therapies to re-train sensory function. The investigators propose to evaluate a novel non-invasive brain stimulation treatment called repetitive Transcranial Magnetic Stimulation (rTMS). The effects of this technique on motor deficits following stroke have been studied, however rTMS for the treatment of sensory loss has not been examined to date. The investigators' study will examine for the first time if rTMS of a sensory brain region can improve sensory function in chronic stroke survivors.

DETAILED DESCRIPTION:
Sensory deficits are present in the majority of stroke survivors. Inability to feel movement, touch or pain impairs the investigators' ability to interact with environment and diminished the quality of life. These sensory deficits significantly impair functional activity and slow down recovery during rehabilitation. Currently available sensory rehabilitation techniques can only partially restore sensory function. The main objective of this study is to test a novel approach to improve sensory function after stroke using non-invasive brain stimulation. This pilot study will measure an immediate effect of different repetitive Transcranial Magnetic Stimulation (rTMS) paradigms in a crossover single session design. The effect of intervention is measured with clinical measures of sensory and motor function and with neurophysiological assessment of sensory pathways. If the concept is demonstrated in this pilot study, then following the lead of other investigations of this type, this pilot will provide the foundation to test the efficacy of a long-term multi-session intervention of combined rTMS and peripherally directed therapy.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable at least 6 months after first ever stroke.
* Sufficient endurance to participate in the study.
* Cognition sufficiently intact to give valid informed consent to participate.
* Age > 18years.
* Ability to follow 2 stage commands.
* Impaired but not absent ability to feel touch, vibration and movement of the affected arm.

Exclusion Criteria:

* Acute or progressive cardiac, renal, respiratory, neurological disorders or malignancy.
* Any psychiatric diagnosis or active psychological condition.
* History of substance abuse within the last 6 months
* More than one ischemic stroke or stroke affecting both sides.
* Claustrophobia, or inability to operate the MRI patient call button.
* Pregnancy or pregnancy planning during the study period.
* Lower motor neuron damage or radiculopathy
* Contraindications for rTMS according to the TMS-use guidelines (Rossi et al 2009).
* Inability to understand English.
* Significant neglect for those with left-sided deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04-12 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Pundik, MD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pundik S, Skelly M, McCabe J, Akbari H, Tatsuoka C, Plow EB. Does rTMS Targeting Contralesional S1 Enhance Upper Limb Somatosensory Function in Chronic Stroke? A Proof-of-Principle Study. Neurorehabil Neural Repair. 2021 Mar;35(3):233-246. doi: 10.1177/1545968321989338. Epub 2021 Jan 29. PMID 33514270

RESULTS

PARTICIPANT FLOW:
Groups:
- Stroke Cohort: Each subject is provided with three different brain stimulation interventions in a single arm, single session crossover design study
  repetitive transcranial magnetic stimulation (rTMS): 3 types of interventions on different sessions
  * session 1 - High frequency rTMS targeting contralesional sensory cortex
  * session 2 - Low frequency rTMS
  * session 3 - sham rTMS
  peripheral sensory stimulation: peripheral sensory electrical stimulation and vibration of the stroke-affected hand administered concurrently with each rTMS
Period: Overall Study
Arm/Group | Stroke Cohort
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Stroke Cohort
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
two point discrimination [Mean (Standard Deviation); unit: mm] — Two-point discrimination was measured with Disk-Criminator disks (Baltimore, MD) by determining the subjects' ability to perceive two points on the disk as two separate points rather than as a single point. The distances between the two points ranged between 2 and 15 mm. One and two sensory points were presented in a pseudo-random order to subjects' 4th digit volar fingertip surface. A threshold is determined when seventy percent accuracy is exhibited for identifying the difference between single versus double point stimulation.
  mm | 12.5 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Two-point Discrimination
Description: Baseline measure is collected immediately before the intervention. There are two data collections following each intervention, one datacollection is immediately after the intervention and the second one is at 1 hour after intervention.
  Two-point discrimination was measured with Disk-Criminator disks (Baltimore, MD) by determining the subjects' ability to perceive two points on the disk as two separate points rather than as a single point. The distances between the two points ranged between 2 and 15 mm. One and two sensory points were presented in a pseudo-random order to subjects' 4th digit volar fingertip surface. A threshold is determined when seventy percent accuracy is exhibited for identifying the difference between single versus double point stimulation.
Time Frame: up to 1 hour after intervention
Population: stroke cohort
Measure: Mean (Standard Deviation); unit: mm
Groups:
- High Frequency rTMS: Each subject is provided with three different brain stimulation interventions in a single arm, single session crossover design study
  For these sessions, participants received 5Hz rTMS targeting contralesional sensory cortex and peripheral sensory stimulation: peripheral sensory electrical stimulation and vibration of the stroke-affected hand administered concurrently with each rTMS
- Low Frequency rTMS: Each subject is provided with three different brain stimulation interventions in a single arm, single session crossover design study
  For these sessions, participants received 1Hz rTMS targeting contralesional sensory cortex and peripheral sensory stimulation: peripheral sensory electrical stimulation and vibration of the stroke-affected hand administered concurrently with each rTMS
- Sham rTMS: Each subject is provided with three different brain stimulation interventions in a single arm, single session crossover design study
  For these sessions, participants received sham Hz rTMS targeting contralesional sensory cortex and peripheral sensory stimulation: peripheral sensory electrical stimulation and vibration of the stroke-affected hand administered concurrently with each rTMS
Arm/Group | High Frequency rTMS | Low Frequency rTMS | Sham rTMS
Number analyzed (Participants) | 16 | 16 | 16
mm
  Immediately post-intervention | -0.7 (2.7) | -0.5 (1.8) | -0.1 (1.3)
  One hour post-intervention | -1.7 (3.5) | -0.3 (1.2) | 0.1 (2.1)

2. Primary Outcome: Change From Baseline in N20 Somatosensory Evoked Potential(SSEP) Peak Latency
Description: Baseline measure is collected immediately before the intervention. Following each intervention, data is collected immediately after each intervention and at 1 hour after intervention.
  SEPs were recorded with a Cadwell Sierra Wave (Cadwell, Kennewick, WA) (LSCDVAMC) or with Powerlab 4/25T (AD Instruments Inc. Colorado Springs, CO) and a Grass Stimulator (Natus Neurology, Middleton, WI) (CC)44. The recording electrodes (1 cm diameter, gold cup electrodes filled with conductive paste) were placed 2 cm posterior to C3 & C4 (10-20 international system of EEG electrode placement) and the reference electrode at Fz (Figure 1). Stimulus was applied to the median nerve at the wrist. Ground electrodes were placed at the lateral epicondyle of the stimulated arm. The evoked response from 500 stimuli were recorded and averaged for a single trial. Three SEP trials were recorded then analyzed. Latencies (in milliseconds) were determined for N20.
Time Frame: up to 1 hour after intervention
Population: stroke cohort
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Sham rTMS: Each subject is provided with three different brain stimulation interventions in a single arm, single session crossover design study
  For these sessions, participants received sham rTMS targeting contralesional sensory cortex and peripheral sensory stimulation: peripheral sensory electrical stimulation and vibration of the stroke-affected hand administered concurrently with each rTMS
Arm/Group | High Frequency rTMS | Low Frequency rTMS | Sham rTMS
Number analyzed (Participants) | 16 | 16 | 16
msec
  Immediately post-intervention | -1.1 (2.3) | 0.1 (2.2) | 0.7 (3.0)
  One hour post-intervention | 0.1 (2.0) | -1.8 (5.8) | 1.2 (2.5)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | High Frequency rTMS | Low Frequency rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT02811913/Prot_SAP_000.pdf